CLINICAL TRIAL: NCT02779634
Title: The Effect of Ubiquinol Treatment on Cardiac Function in Patients With Heart Failure With Preserved Ejection Fraction
Brief Title: Ubiquinol Treatment in Patients With Heart Failure and Preserved Ejection Fraction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, LEIBOWITZ DAVID, Associate professor of medicine Hadassah-Hebrew University Medical Center, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COENZYMEQ
Record Dates: First submitted 2016-05-15; First posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — ubiquinol; coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo three times daily
  Interventions: Drug: Placebo
- Active (Active Comparator): Pills of 100 mg ubiquinol three times daily
  Interventions: Drug: ubiquinol

INTERVENTIONS:
Drug: ubiquinol — Ubiquinol three times daily
  Other Names: coenzyme Q10
  Arms: Active
Drug: Placebo — Sugar pill three times daily
  Arms: Placebo

SUMMARY:
There are no studies specifically examining the effects of coenzyme Q (CoQ) treatment on echocardiographic indices of diastolic function in elderly patients with heart failure with preserved ejection fraction (HFPEF). In previous studies the only echocardiographic parameters studied were ejection fraction (EF) and chamber size. The objective of the proposed current study is to examine the effect of 16 weeks of ubiquinol therapy on diastolic function assessed by echocardiography in patients over the age of 50 with a clinical diagnosis of HFPEF. Ubiquinol (Kaneka Pharma), the reduced form of CoQ will be utilized for this study as it has been shown to have superior bioavailability when compared to oxidized CoQ.

ELIGIBILITY:
Inclusion Criteria:

* Typical signs and symptoms of congestive heart failure (CHF) (New York Association Class 2-4).
* Normal ejection fraction on echocardiography (EF ≥50%).
* Evidence of diastolic dysfunction on non-invasive imaging (E:e' > 15 or e:e' > 8 with other measures of diastolic dysfunction such as e/a < 0.5 with elevated deceleration time or left atrial volume index > 40 cc/m2 or presence of elevated left ventricular mass index or elevated pulmonary pressures).
* Stable medical therapy for 4 weeks prior to randomization

Exclusion Criteria:

* Chronic atrial fibrillation.
* Acute coronary syndrome or coronary revascularization within 60 days.
* Clinically significant valvular disease.
* Known infiltrative cardiomyopathy (e.g. amyloidosis), hypertrophic cardiomyopathy or chronic pericardial disease.
* Inability/refusal to provide informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change in diastolic function as assessed by mitral valve inflow and tissue Doppler velocities on echocardiography | 4 months
NT-pro brain natriuretic peptide (NT-proBNP) serum levels (pg/ml) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: David Leibowitz, MD, Principal Investigator — Hadassah Medical Organization

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Samuel TY, Hasin T, Gotsman I, Weitzman T, Ben Ivgi F, Dadon Z, Asher E, Amir O, Glikson M, Alcalai R, Leibowitz D. Coenzyme Q10 in the Treatment of Heart Failure with Preserved Ejection Fraction: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial. Drugs R D. 2022 Mar;22(1):25-33. doi: 10.1007/s40268-021-00372-1. Epub 2021 Nov 26. PMID 34826125